CLINICAL TRIAL: NCT04160585
Title: Musculoskeletal Pain Among Turkish Office Workers
Brief Title: Individual and Work-Related Risk Factors for Musculoskeletal Pain: a Cross-Sectional Study Among Turkish Office Workers
Status: Completed | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Tansu Birinci, PT, MSc Research Assistant, Istanbul University - Cerrahpasa
Other Study IDs: 10112019
Record Dates: First submitted 2019-11-09; First posted 2019-11-13 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Musculoskeletal Pain; Disability Physical
MeSH Terms: conditions — Musculoskeletal Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: There is no intervention. — There is no intervention.

SUMMARY:
Most studies investigating the risk factors related with musculoskeletal pain have been conducted in European countries and North America, and because of the difference in health, economic, and social systems, their results are not generalizable to countries such as Turkey. Therefore, the aim of the present study is to investigate the individual and work-related risk factors linked to musculoskeletal pain among Turkish office workers.

DETAILED DESCRIPTION:
A total of 150 participants, who are office workers in Turkey, are included in the present study. Data collection will be carried out using the online survey. The online survey link will be shared via social media accounts and via mail. The questionnaire created through Google forms will be delivered to the participants via the link. The link will be active in the data collection process. Before the participants start the questionnaire, they will be asked whether they were willing to participate. The socio-demographic characteristics (age, gender, body mass index) and health status (presence of chronic disease, drugs used and history of injury) will be questioned. In addition, the information about the sector, working hours, time spent at work and out of work, additional working hours, break times at the workplace will be collected. The Standardized Scandinavian Musculoskeletal Questionnaire will be used to assess musculoskeletal complaints. Participants with musculoskeletal pain will be referred to the assessment questionnaire appropriate for the localization of the region where they feel the most pain. Participants with neck pain will be evaluated with the Neck Disability Scale. Arm-Shoulder-Hand Disability Survey-Short Form will be used for participants with wrist, shoulder or arm pain. Oswestry Disability Index will be used to determine the degree of disability in individuals with low back pain.

ELIGIBILITY:
Inclusion Criteria:

* The participants included in this study will be aged between 18 and 55 years, men or women, an office worker and able to understand and read Turkish as a language.

Exclusion Criteria:

* Participants excluded from the study if they have any musculoskeletal disease, a spine curvature disorders such as scoliosis, kyphosis, kyphoscoliosis, undergone surgery affecting the musculoskeletal system within the last 1 month, or been pregnant for women.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: A total of 150 participants, who are office workers in Turkey, will be included in the present study.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
The Standardized Scandinavian Musculoskeletal Questionnaire | Baseline
  The Standardized Scandinavian Musculoskeletal Questionnaire (NMQ) will be used to assess musculoskeletal complaints. NMQ is a questionnaire that evaluates wrist, neck, shoulder and general musculoskeletal complaints with standardized questions. In NMQ; pain and discomfort are questioned in the last 12 months and the last seven days, the mapping of the body in specific nine regions (feet-ankles, knees, thighs, hips, ankles, hands, waist, elbows, back, shoulders, neck) and whether this situation interferes with the usual work. At the end of the NMQ, the participants are encountered by the question of "Do you have any pain related to the musculoskeletal system? and Which region is the most painful?" Surveys of participants who do not feel any pain due to the musculoskeletal system were completed.

SECONDARY OUTCOMES:
Neck Disability Scale | Baseline
  The Neck Disability Scale is based on the Oswestry Low Back Pain Disability Index and consists of 10 topics. Pain sensitivity includes personal care, weight lifting, reading, headaches, concentration, work/work, driving, sleep, and social activities. Each question has 6 response options that measure the severity of pain or limitation Scoring is done between 0-5 and the total score is calculated between 0-50. According to the total score, there is no limitation between 0-4 points; Slight limitation of 5-14; Moderate limitation of 15-24; Serious limitations between 25-34; 34 and above are classified as totally restricted.
Arm-Shoulder-Hand Disability Survey-Short Form | Baseline
  Arm-Shoulder-Hand Disability Survey-Short Form (Quick DASH, Q-DASH) will be used for participants with wrist, shoulder or arm pain. Q-DASH is a regional outcome measure developed for upper extremity musculoskeletal disorders and should include 11 questions, at least 10 of 11 questions should be answered in order to calculate the score of the scale reported to be used instead of DASH. Each question is scored on a 5-point scale and a final score ranging from 0 (no disability) to 100 (severe disability) is calculated.
Oswestry Disability Index | Baseline
  Oswestry Disability Index (ODI) will be used to determine the degree of disability in individuals with low back pain. ODI consists of a total of 10 items measuring the severity of pain, personal care, lifting, walking, sitting, standing, social life, sleep, travel and pain. Each item is rated between 0-5. As the total score increases, the level of disability increases. The maximum score is 50 points; It is evaluated as severe between 31-50 points, moderate between 11-30 points and mild between 1-10 points. The total score obtained from the patient can be converted to the percentage system and calculated as a percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Tansu Birinci, MSc, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Bakırkoy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No